CLINICAL TRIAL: NCT05077085
Title: New Treatment Strategy for Patients With Multiple Recurrent Clostridioides Difficile Infection With Bezlotoxumab as First Option
Brief Title: Bezlotoxumab Versus FMT for Multiple Recurrent CDI
Acronym: BSTEP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Leiden University Medical Center (Other)
Collaborators: OLVG (Network); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, Joffrey van Prehn, MD, PhD, Clinical Microbiologist, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSTEP
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Clostridium Infections; Clostridioides Difficile; Enterocolitis, Pseudomembranous
MeSH Terms: conditions — Clostridium Infections; Enterocolitis, Pseudomembranous | interventions — bezlotoxumab; Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Intervention Model Description: Multicenter open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strategy A: initial SoC + bezlotoxumab. SoC + FMT rescue therapy. (Experimental): initial bezlotoxumab in addition to 14 days SoC oral antibiotic treatment with vancomycin 125 mg QID. 14 days of vancomycin 125mg QID plus fecal microbiota in case of treatment failure.
  Interventions: Drug: Bezlotoxumab; Drug: Vancomycin oral
- Strategy B: initial SoC + FMT. Fidaxomicin rescue therapy. (Active Comparator): fecal microbiota transplantation in addition to 14 days SoC oral antibiotic treatment with vancomycin 125 mg QID. 10 days of fidaxomicin 200 mg BID in case of treatment failure.
  Interventions: Procedure: Fecal Microbiota Transplantation (FMT); Drug: Vancomycin oral

INTERVENTIONS:
Drug: Bezlotoxumab — single intravenous infusion of bezlotoxumab 10 mg/kg
  Arms: Strategy A: initial SoC + bezlotoxumab. SoC + FMT rescue therapy.
Procedure: Fecal Microbiota Transplantation (FMT) — single infusion of 198 cc fecal suspension (derived from 60g donor feces) via duodenal tube or coloscopy
  Arms: Strategy B: initial SoC + FMT. Fidaxomicin rescue therapy.
Drug: Vancomycin oral — 14 days vancomycin oral 125mg QID (250mg QID when 125mg not available)

SUMMARY:
The objective of this trial is to investigate whether a treatment strategy offering bezlotoxumab before FMT in patients suffering from multiple recurrent CDI results in equal efficacy compared with a treatment strategy with initial FMT. Strategy A includes bezlotoxumab as ancillary treatment as first option, and FMT in case of failure. Option B includes FMT as ancillary treatment as first option, and antibiotic treatment with fidaxomicin in case of failure. A secondary objective is to provide a point estimate of recurrence after bezlotoxumab for the treatment of multiple recurrent CDI.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* diarrhea (3 or more unformed stools per 24h for two consecutive days; or >= 8 unformed stools per 48h) XML File Identifier: KqQEbBLRYEZjGgsIl5GcI+NXCyM= Page 10/22
* positive PCR test for toxin A/B genes and/or positive toxin EIA for current and previous episodes (low PCR cycle threshold value when only PCR performed)
* a minimum of two prior CDI episodes
* previous episode is maximum of 3 months prior to the current episode
* the current episode responds well to Standard of Care treatment (vancomycin or fidaxomicin orally).
* Assessment of the severity of the disease will be performed according to the ESCMID recommendations.
* Both mild and severe CDI will be included

Exclusion Criteria:

* Severe complicated CDI, i.e presence of: hypotension, septic shock, elevated serum lactate, ileus, toxic megacolon, bowel perforation, or any fulminant course of disease.
* ICU admission for underlying disease
* pregnancy or current desire for pregnancy
* breastfeeding
* (prolonged) use of antibiotics (other than for treatment of CDI) during the study period or directly after the intervention
* previous use of bezlotoxumab or fecal microbiota transplantation
* a history of underlying congestive heart failure (potential safety signal phase-III trail bezlotoxumab).
* Diagnosis of inflammatory bowel disease in medical history.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Global cure of the treatment strategy | 12 weeks (after rescue therapy if applicable)
  Defined as cure without relapse of CDI within 12 weeks after completion of the treatment strategy in the study arm, i.e. after completion of secondary treatment in case of failure on initial treatment.

SECONDARY OUTCOMES:
Initial cure after treatment with bezlotoxumab or FMT | 2 days after end of treatment
  Defined as cure after completion of the primary CDI treatment in the study arm. Initial cure is assessed at day 2 after end of treatment (EOT).
Recurrence after initial treatment with bezlotoxumab or FMT | 12 weeks
  Defined as CDI relapse within 12 weeks after initial cure
Sustained cure after initial treatment with bezlotoxumab or FMT | 12 weeks
  Sustained cure is defined as cure without relapse of CDI within 12 weeks after completion of the initial treatment.
Adverse events | 12 weeks
  Throughout the entire study all adverse events will be noted. After the final study procedure of the last patient, all adverse events will be categorized:
  1. Most likely related to ancillary CDI treatment (bezlotoxumab or FMT)
  2. May be related to ancillary CDI treatment
  3. Not related to ancillary CDI treatment
Post-treatment IBS-like symptoms | 12 weeks
  Development of post-treatment irritable bowel syndrome like symptoms associated with bezlotoxumab treatment or FMT treatment
Duration of hospitalization | 12 weeks
Rate of antibiotic use | 12 weeks
Eradication of toxigenic C. difficile | 3 and 12 weeks
  As assessed by PCR
Fecal microbiota (16S) alfa- and beta-diversity | Pre-treatment and 3 and 12 weeks
  As assessed by 16S rRNA amplicon sequencing
Cost-effectiveness | 12 weeks
  Costs per cured patient (global and sustained cure) and costs per QALY gained, using the EQ-5D-5L health questionaire that assesses five domains by 5 point scale, e.g. no/slight/moderate/severe/extreme impairment and a visual analogue 0-100 scale of health rating, higher is better)

OTHER OUTCOMES:
Patient wellbeing | Pre-treatment and 12 weeks
  As assessed by questionnaire, that includes:
  1. self rated health - 5 point scale, higher is worse outcome
  2. happiness - 7 points scale, higher is worse outcome
  3. optimism - 6 items
  4. patient health questionnaire PHQ-9 - 9 items with 4 point scale, higher is worse outcome
  5. hospital anxiety and depression scale HADS - 14 items
Rate of patients with improved defecation pattern | 12 weeks
  As assessed by personal diary

CONTACTS AND LOCATIONS:
Overall Officials: J van Prehn, Principal Investigator — Leiden University Medical Center
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Centers, AMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medical Center, The Hague

IPD SHARING:
Plan to Share IPD: No